CLINICAL TRIAL: NCT00312858
Title: An Open, Randomized, Multicenter Study of the Safety, Tolerability, & Immunogenicity of VAQTA™ Given Concomitantly With PROQUAD™ and PREVNAR™ in Healthy Children 12 Months of Age
Brief Title: Concomitant Use of Hepatitis A Vaccine With Measles, Mumps, Rubella and Varicella Vaccine and Pneumococcal 7-Valent Conjugate Vaccine in Healthy 12-Month-Old Children (V251-067)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V251-067; 2005_075
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis A Virus
Keywords: Hepatitis A Virus
MeSH Terms: conditions — Hepatitis | interventions — Hepatitis A Vaccines; Chickenpox Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Arm 1: VAQTA™ 0.5 mL injection (2 doses 6 months apart), ProQuad™ 0.5 mL injection (2 doses 6 months apart), Prevnar™ 0.5 mL injection (one dose), all vaccines administered concomitantly. 28 weeks of study duration.
  Interventions: Biological: Comparator: VAQTA™ (Hepatitis A vaccine); Biological: Comparator: ProQuad™ (Measles, Mumps, Rubella and Varicella vaccine); Biological: Comparator: Prevnar™ (Pneumococcal 7-Valent Conjugate vaccine)
- 2 (Active Comparator): Arm 2: ProQuad™ 0.5 mL injection (2 doses ~8 months apart), Prevnar™ 0.5 mL injection (one dose), both administered concomitantly, VAQTA™ 0.5 mL injection (2 doses 6 months apart) administered alone. 34 weeks of study duration.
  Interventions: Biological: Comparator: VAQTA™ (Hepatitis A vaccine); Biological: Comparator: ProQuad™ (Measles, Mumps, Rubella and Varicella vaccine); Biological: Comparator: Prevnar™ (Pneumococcal 7-Valent Conjugate vaccine)

INTERVENTIONS:
Biological: Comparator: VAQTA™ (Hepatitis A vaccine) — VAQTA™ 0.5 mL injection
Biological: Comparator: ProQuad™ (Measles, Mumps, Rubella and Varicella vaccine) — ProQuad™ 0.5 mL injection
Biological: Comparator: Prevnar™ (Pneumococcal 7-Valent Conjugate vaccine) — Prevnar™ 0.5 mL injection

SUMMARY:
Hepatitis A vaccine will be given either alone or together with measles, mumps, rubella, and varicella vaccine and pneumococcal 7-valent conjugate vaccine at the first dose and together with measles, mumps, rubella, and varicella [Oka/Merck] virus vaccine at the second dose. Immunogenicity and safety data will be collected after each dose of vaccine.

DETAILED DESCRIPTION:
Vaccines: V251, Hepatitis A Vaccine, Inactivated (VAQTA™) administered with Measles, Mumps, Rubella and Varicella Vaccine (ProQuad™) and Pneumococcal 7-Valent Conjugate Vaccine (Prevnar™) will have a Duration of Treatment: 2 Doses, 6 months apart.

Vaccine: Hepatitis A Vaccine, Inactivated (VAQTA™), administered alone will have a Duration of Treatment: 2 Doses, 6 months apart.

ELIGIBILITY:
Inclusion Criteria:

* 12- to 15-month-old males and females with no active liver disease
* A negative history of hepatitis A, measles, mumps, rubella, chickenpox, and/or zoster

Exclusion Criteria:

* Males and females previously vaccinated with hepatitis A, measles, mumps, rubella, and/or chickenpox vaccine
* Any immune deficiency
* History of allergy to any of the vaccine components
* History of any seizure disorder

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 653 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Yetman RJ, Shepard JS, Duke A, Stek JE, Petrecz M, Klopfer SO, Kuter BJ, Schodel FP, Lee AW. Concomitant administration of hepatitis A vaccine with measles/mumps/rubella/varicella and pneumococcal vaccines in healthy 12- to 23-month-old children. Hum Vaccin Immunother. 2013 Aug;9(8):1691-7. doi: 10.4161/hv.24873. Epub 2013 Jun 6. PMID 23744509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 clinical sites in the United States
  Date first participant visit: 14-Apr-2006
  Date last participant visit: 25-Mar-2008
Groups:
- Arm 1: VAQTA™ + ProQuad™ + Prevnar™: VAQTA™ (hepatitis A vaccine) + ProQuad™ (measles, mumps, rubella, and varicella vaccine) + Prevnar™ (pneumococcal 7-valent conjugate vaccine) administered at the same time at first study visit. Second doses of VAQTA™ and ProQuad™ administered together 24 weeks later at third study visit.
- Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™: VAQTA™ (hepatitis A vaccine) dose 1 administered separately from ProQuad™ (measles, mumps, rubella, and varicella vaccine) and Prevnar™ (pneumococcal 7-valent conjugate vaccine). A second dose of VAQTA™ administered 24 weeks after the first dose at third study visit.
Period: Overall Study
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Started | 330 | 323
Visit 1 | 330 | 323
Visit 2 | 305 | 294
Visit 3 | 273 | 261
Visit 4 | 262 | 240
Completed | 262 | 230
Not Completed | 68 | 93
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 25 | 42
Not completed — Protocol Violation | 3 | 8
Not completed — Withdraw by Participant | 20 | 20
Not completed — Participant Moved | 11 | 10
Not completed — Other | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™ | Total
Number analyzed (Participants) | 330 | 323 | 653
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.4 (0.80) | 12.5 (0.89) | 12.4 (0.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 166 | 322
  Male | 174 | 157 | 331

OUTCOME MEASURES:

1. Primary Outcome: Antibody Response to Hepatitis A - Participants With a Serological Response
Description: Number of participants with titer ≥10 mIU/mL, i.e., seropositive for hepatitis A antibody, regardless of initial serostatus
Time Frame: 4 weeks Postdose 2 of hepatitis A vaccine (VAQTA™)
Population: Per-protocol analysis set includes participants who received 2 doses of VAQTA™ (hepatitis A vaccine), had a Postdose 2 serology results, and followed the protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 182 | 159
Participants | 182 | 158
Statistical Analysis 1: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Comparison of the difference (percentage points) in estimated response rates of Arm 1 - Arm 2; Test type: Non-Inferiority or Equivalence — Similarity (non-inferiority) based on lower bound of the 2-sided 95% CI on the risk difference of seroresponse rates excluding a decrease of 10 percentage points or more (lower bound >-10.0); p < 0.001, Miettinen and Nurminen — Similarity (non-inferiority) indicated that the risk difference was statistically significantly greater than the pre-specified clinically relevant difference of -10 percentage points at the 1-sided α=0.025 level; For testing the non-inferiority of 2 proportions. Stratified by investigator; Risk Difference (RD) = 0.7, 95% CI [-1.4 to 3.8] — Difference in estimated response rates of Arm 1 - Arm 2

2. Primary Outcome: Antibody Response to Varicella - Participants With a Serological Response
Description: Participants with varicella baseline antibody titer <1.25 gpELISA units/mL and Postdose 1 titers ≥1.25 gpELISA units/mL (seroconversion) and ≥5 gpELISA units/mL (seroprotection)
Time Frame: 6 weeks Postdose 1 of varicella-containing vaccine (ProQuad™)
Population: Per-protocol analysis set includes participants who received the initial dose of ProQuad™ (varicella-containing vaccine), had a Postdose 1 serology result, and followed the protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 225 | 232
Participants
  Number of participants ≥1.25 gpELISA units/mL | 222 | 231
  Number of participants ≥5 gpELISA units/mL | 210 | 228
Statistical Analysis 1: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Comparison of the difference (percentage points) in estimated response rates of Arm 1 - Arm 2 for participants with initial serostatus <1.25 gpELISA units/mL; Test type: Non-Inferiority or Equivalence — Similarity (non-inferiority) based on lower bound of the 2-sided 95% CI on the risk difference seroresponse rates excluding a decrease of 10 percentage points or more (lower bound >-10.0); p = 0.013, Miettinen and Nurminen — Similarity (non-inferiority) indicated that the risk difference was statistically significantly greater than the pre-specified clinically relevant difference of -10 percentage points at the 1-sided multiplicity-adjusted α=0.025 level; For testing the non-inferiority of 2 proportions. Stratified by investigator; Risk Difference (RD) = -5.1, 95% CI [-9.3 to -1.4] — Difference in estimated response rates of Arm 1 - Arm 2

3. Primary Outcome: Antibody Response to Streptococcus Pneumoniae - Geometric Mean Titers
Description: Serum antibodies to serotype-specific pneumococcal polysaccharides were determined by enzyme-linked immunosorbent assay
Time Frame: 6 weeks Postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 330 | 323
mcg/mL
  Serotype 4 (n=246, 247) | 1.8 [1.6 to 2.1] | 1.6 [1.4 to 1.8]
  Serotype 6B (n=246, 246) | 9.5 [8.3 to 11.0] | 9.6 [8.5 to 10.8]
  Serotype 9V (n=247, 247) | 3.7 [3.2 to 4.2] | 4.1 [3.7 to 4.7]
  Serotype 14 (n=248, 247) | 7.7 [6.8 to 8.8] | 7.4 [6.5 to 8.4]
  Serotype 18C (n=247, 247) | 2.9 [2.6 to 3.3] | 2.6 [2.3 to 3.0]
  Serotype 19F (n=248, 248) | 4.0 [3.5 to 4.5] | 3.8 [3.3 to 4.3]
  Serotype 23F (n=247, 247) | 4.9 [4.3 to 5.6] | 4.5 [3.9 to 5.1]
Statistical Analysis 1: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Serotype 4; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion is met if the lower bound of the 95% confidence interval of the response ratio is >0.5, excluding a decrease of 2-fold or more; p < 0.001, ANCOVA; Response ratio (Arm 1 / Arm 2) = 1.1, 95% CI 2-sided [0.9 to 1.3] — Response ratio is based on statistical models adjusting the GMT for combined study center and prevaccination titer
Statistical Analysis 2: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Response ratio (Arm 1 / Arm 2) = 1.0, 95% CI 2-sided [0.8 to 1.2] — Response ratio is based on statistical models adjusting the GMT for combined study center and prevaccination titer
Statistical Analysis 3: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Response ratio (Arm 1 / Arm 2) = 0.9, 95% CI 2-sided [0.8 to 1.0] — Response ratio is based on statistical models adjusting the GMT for combined study center and prevaccination titer
Statistical Analysis 4: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Response ratio (Arm 1 / Arm 2) = 1.0, 95% CI 2-sided [0.9 to 1.2] — Response ratio is based on statistical models adjusting the GMT for combined study center and prevaccination titer
Statistical Analysis 5: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Response ratio (Arm 1 / Arm 2) = 1.1, 95% CI 2-sided [0.9 to 1.3] — Response ratio is based on statistical models adjusting the GMT for combined study center and prevaccination titer
Statistical Analysis 6: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Response ratio (Arm 1 / Arm 2) = 1.1, 95% CI 2-sided [0.9 to 1.2] — Response ratio is based on statistical models adjusting the GMT for combined study center and prevaccination titer
Statistical Analysis 7: Comparison: Arm 1: VAQTA™ + ProQuad™ + Prevnar™ vs Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™; Serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Response ratio (Arm 1 / Arm 2) = 1.1, 95% CI 2-sided [1.0 to 1.3] — Response ratio is based on statistical models adjusting the GMT for combined study center and prevaccination titer

4. Primary Outcome: Participants With 1 or More Systemic Adverse Experience
Description: Systemic adverse experiences are unfavorable or unintended changes in the body after getting study vaccine. They are collected the first 14 days after receipt of dose 1 of hepatitis A vaccine (VAQTA™) (Days 1 to 14) within the 6 week study period.
Time Frame: 6 weeks post dose 1
Population: Includes all participants who provided safety follow-up after receipt of Dose 1 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 311 | 274
Participants | 178 | 80

5. Primary Outcome: Participants With 1 or More Systemic Adverse Experience
Description: Systemic adverse experiences are unfavorable or unintended changes in the body after getting study vaccine. They are collected the first 14 days after receipt of dose 2 of hepatitis A vaccine (VAQTA™) (Days 1 to 14) within the 4 week study period.
Time Frame: 4 weeks post dose 2
Population: Includes all participants who provided safety follow-up after receipt of Dose 2 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 263 | 251
Participants | 88 | 77

6. Primary Outcome: Participants With 1 or More Systemic Adverse Experience.
Description: Systemic adverse experiences are unfavorable or unintended changes in the body after getting study vaccine. Collected the first 14 days after each of the 2 doses of hepatitis A vaccine (VAQTA™) (Days 1 to 14), given 6 months apart
Time Frame: 6 months
Population: Includes all participants who provided safety follow-up after receipt of any dose of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 330 | 286
Participants | 204 | 133

7. Primary Outcome: Participants With 1 or More Injection-site Adverse Experience
Description: Injection-site adverse experiences collected the first 5 days after receipt of dose 1 of hepatitis A vaccine (VAQTA™) (Days 1 to 5) within the 6 week study period.
Time Frame: 6 weeks post dose 1
Population: Includes all participants who provided safety follow-up after receipt of Dose 1 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 311 | 274
Participants | 83 | 61

8. Primary Outcome: Participants With 1 or More Injection-site Adverse Experience
Description: Injection-site adverse experiences collected the first 5 days after receipt of dose 2 of hepatitis A vaccine (VAQTA™) (Days 1 to 5) within the 4 week study period.
Time Frame: 4 weeks post dose 2
Population: Includes all participants who provided safety follow-up after receipt of Dose 2 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 263 | 251
Participants | 54 | 66

9. Primary Outcome: Participants With 1 or More Injection-site Adverse Experience
Description: Injection-site adverse experiences collected the first 5 days after receipt of each dose of hepatitis A vaccine (VAQTA™) (Days 1 to 5) over the 6 months in which the 2 doses of vaccine were administered.
Time Frame: 6 months
Population: Includes all participants who provided safety follow-up after receipt of any dose of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 330 | 286
Participants | 105 | 95

10. Primary Outcome: Participants With Elevated Temperature (≥102.2F/ ≥39.0C)
Description: Elevated temperatures measured the first 5 days after receipt of dose 1 of hepatitis A vaccine (VAQTA™) (Days 1 to 5) within the 6 week study period.
Time Frame: 6 weeks post dose 1
Population: Includes all participants who provided safety follow-up after receipt of Dose 1 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 285 | 243
Participants | 10 | 5

11. Primary Outcome: Participants With Elevated Temperature (≥102.2F/ ≥39.0C)
Description: Elevated temperatures measured the first 5 days after receipt of dose 2 of hepatitis A vaccine (VAQTA™) (Days 1 to 5) within the 4 week study period.
Time Frame: 4 weeks post dose 2
Population: Includes all participants who provided safety follow-up after receipt of Dose 2 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 237 | 221
Participants | 6 | 5

12. Primary Outcome: Participants With Elevated Temperature (≥102.2F/ ≥39.0C)
Description: Elevated temperatures measured the first 5 days after receipt of each dose of hepatitis A vaccine (VAQTA™) (Days 1 to 5) over the 6 months in which the 2 doses of vaccine were administered.
Time Frame: 6 months
Population: Includes all participants who provided safety follow-up after receipt of any dose of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 293 | 257
Participants | 16 | 10

13. Primary Outcome: Participants With 1 or More Serious Vaccine-related Adverse Experience
Description: Serious vaccine-related adverse experience causes death, persistent or significant disability, causes or prolong a hospital stay, is a cancer, an overdose, or life-threatening. They were collected during the entire study and believed due to study vaccine
Time Frame: 6 weeks post dose 1
Population: Includes all participants who provided safety follow-up after receipt of Dose 1 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 311 | 274
Participants | 0 | 1

14. Primary Outcome: Participants With 1 or More Serious Vaccine-related Adverse Experience
Description: as for outcome 13
Time Frame: 4 weeks post dose 2
Population: Includes all participants who provided safety follow-up after receipt of Dose 2 of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 263 | 251
Participants | 0 | 0

15. Primary Outcome: Participants With 1 or More Serious Vaccine-related Adverse Experience
Description: as for outcome 13
Time Frame: 6 months
Population: Includes all participants who provided safety follow-up after receipt of any dose of VAQTA™ (hepatitis A vaccine)
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 330 | 286
Participants | 0 | 1

16. Other Pre Specified Outcome: Antibody Response to Hepatitis A - Geometric Mean Titer
Description: Geometric Mean Titer of hepatitis A antibody, regardless of initial serostatus
Time Frame: 4 weeks Postdose 2 of hepatitis A vaccine (VAQTA™)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 182 | 159
mIU/mL | 4976.6 [4067.6 to 6088.6] | 6123.2 [4825.6 to 7769.7]

17. Other Pre Specified Outcome: Antibody Response to Varicella - Geometric Mean Titer
Description: Geometric Mean Titer of varicella antibody, baseline antibody titer was <1.25 gpELISA units/mL
Time Frame: 6 weeks Postdose 1 of varicella-containing vaccine (ProQuad™)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 225 | 232
gpELISA units/mL | 14.6 [13.3 to 16.1] | 16.4 [15.1 to 17.7]

18. Other Pre Specified Outcome: Antibody Response to S. Pneumoniae Serotype 4 - Participants With a Serological Response
Description: Number of participants with a postvaccination titer >=0.2 mcg/mL for S. pneumoniae serotype 4
Time Frame: 6 weeks postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures. Serotype 4 is one of 7 individual serotypes contained in Prevnar™.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 246 | 247
Participants | 241 | 237

19. Other Pre Specified Outcome: Antibody Response to S. Pneumoniae Serotype 6B - Participants With a Serological Response
Description: Number of participants with a postvaccination titer >=0.2 mcg/mL for S. pneumoniae serotype 6B
Time Frame: 6 weeks postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures. Serotype 6B is one of 7 individual serotypes contained in Prevnar™.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 246 | 246
Participants | 242 | 245

20. Other Pre Specified Outcome: Antibody Response to S. Pneumoniae Serotype 9V - Participants With a Serological Response
Description: Number of participants with a postvaccination titer >=0.2 mcg/mL for S. pneumoniae serotype 9V
Time Frame: 6 weeks postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures. Serotype 9V is one of 7 individual serotypes contained in Prevnar™.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 247 | 247
Participants | 243 | 245

21. Other Pre Specified Outcome: Antibody Response to S. Pneumoniae Serotype 14 - Participants With a Serological Response
Description: Number of participants with a postvaccination titer >=0.2 mcg/mL for S. pneumoniae serotype 14
Time Frame: 6 weeks postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures. Serotype 14 is one of 7 individual serotypes contained in Prevnar™.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 248 | 247
Participants | 245 | 244

22. Other Pre Specified Outcome: Antibody Response to S. Pneumoniae Serotype 18C - Participants With a Serological Response
Description: Number of participants with a postvaccination titer >=0.2 mcg/mL for S. pneumoniae serotype 18C
Time Frame: 6 weeks postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures. Serotype 18C is one of 7 individual serotypes contained in Prevnar™.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 247 | 247
Participants | 245 | 243

23. Other Pre Specified Outcome: Antibody Response to S. Pneumoniae Serotype 19F - Participants With a Serological Response
Description: Number of participants with a postvaccination titer >=0.2 mcg/mL for S. pneumoniae serotype 19F
Time Frame: 6 weeks postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures. Serotype 19F is one of 7 individual serotypes contained in Prevnar™.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 248 | 248
Participants | 245 | 244

24. Other Pre Specified Outcome: Antibody Response to S. Pneumoniae Serotype 23F - Participants With a Serological Response
Description: Number of participants with a postvaccination titer >=0.2 mcg/mL for S. pneumoniae serotype 23F
Time Frame: 6 weeks postvaccination of pneumococcal 7-valent conjugate vaccine (Prevnar™)
Population: Per-protocol analysis set includes participants who received Prevnar™ (pneumococcal 7-valent conjugate vaccine), had a postvaccination serology result, and followed the protocol procedures. Serotype 23F is one of 7 individual serotypes contained in Prevnar™.
Measure: Number; unit: Participants
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Number analyzed (Participants) | 247 | 247
Participants | 245 | 246

ADVERSE EVENTS:
Arm/Group | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Serious Adverse Events (participants affected / at risk) | 2 | 6
Other Adverse Events (participants affected / at risk) | 231 | 172
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Pneumonia (Infections and infestations) | 1/330 (1) | 0/323 (0)
Cellulitis (Infections and infestations) | 1/330 (1) | 0/323 (0)
Perineal Abscess (Infections and infestations) | 1/330 (1) | 0/323 (0)
Genital Abscess (Infections and infestations) | 0/330 (0) | 1/323 (1)
Bronchopneumonia (Infections and infestations) | 0/330 (0) | 1/323 (1)
Gastroenteritis (Infections and infestations) | 0/330 (0) | 2/323 (2)
Dehydration (Metabolism and nutrition disorders) | 0/330 (0) | 2/323 (2)
Febrile Convulsion (Nervous system disorders) | 0/330 (0) | 1/323 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0/330 (0) | 1/323 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Arm 1: VAQTA™ + ProQuad™ + Prevnar™ | Arm 2: VAQTA™ Separate From ProQuad™ and Prevnar™
Lymphadenopathy (Blood and lymphatic system disorders) | 1/330 | 0/286
Ear Pain (Ear and labyrinth disorders) | 2/330 | 2/286
Otorrhea (Ear and labyrinth disorders) | 0/330 | 1/286
Conjunctivitis (Eye disorders) | 3/330 | 4/286
Eye Discharge (Eye disorders) | 2/330 | 0/286
Eye Swelling (Eye disorders) | 0/330 | 1/286
Abdominal Pain Upper (Gastrointestinal disorders) | 1/330 | 0/286
Constipation (Gastrointestinal disorders) | 2/330 | 1/286
Diarrhea (Gastrointestinal disorders) | 16/330 | 8/286
Flatulence (Gastrointestinal disorders) | 0/330 | 1/286
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1/330 | 0/286
Nausea (Gastrointestinal disorders) | 0/330 | 1/286
Oral Pain (Gastrointestinal disorders) | 0/330 | 1/286
Teething (Gastrointestinal disorders) | 0/330 | 1/286
Vomiting (Gastrointestinal disorders) | 10/330 | 6/286
Body Temperature (General disorders) | 1/330 | 0/286
Fatigue (General disorders) | 1/330 | 1/286
Irritability (General disorders) | 24/330 | 17/286
Pain (General disorders) | 0/330 | 1/286
Pyrexia (General disorders) | 126/330 | 53/286
Drug Hypersensitivity (Immune system disorders) | 1/330 | 0/286
Multiple Allergies (Immune system disorders) | 3/330 | 0/286
Seasonal Allergy (Immune system disorders) | 0/330 | 1/286
Acute Sinusitis (Infections and infestations) | 1/330 | 0/286
Adenovirus Infection (Infections and infestations) | 0/330 | 1/286
Body Tinea (Infections and infestations) | 1/330 | 0/286
Bronchitis (Infections and infestations) | 1/330 | 1/286
Candida Nappy Rash (Infections and infestations) | 2/330 | 1/286
Candidiasis (Infections and infestations) | 0/330 | 1/286
Conjunctivitis Bacterial (Infections and infestations) | 0/330 | 1/286
Conjunctivitis Infective (Infections and infestations) | 3/330 | 1/286
Conjunctivitis Viral (Infections and infestations) | 1/330 | 0/286
Croup Infectious (Infections and infestations) | 3/330 | 4/286
Ear Infection (Infections and infestations) | 6/330 | 1/286
Enterobiasis (Infections and infestations) | 0/330 | 1/286
Eye Infection (Infections and infestations) | 2/330 | 0/286
Gastroenteritis (Infections and infestations) | 3/330 | 2/286
Gastroenteritis Viral (Infections and infestations) | 2/330 | 3/286
Impetigo (Infections and infestations) | 1/330 | 0/286
Influenza (Infections and infestations) | 1/330 | 2/286
Mycoplasma Infection (Infections and infestations) | 0/330 | 1/286
Nasopharyngitis (Infections and infestations) | 12/330 | 7/286
Otitis Media (Infections and infestations) | 25/330 | 17/286
Otitis Media Acute (Infections and infestations) | 2/330 | 3/286
Pharyngitis (Infections and infestations) | 3/330 | 3/286
Pharyngitis Streptococcal (Infections and infestations) | 2/330 | 3/286
Pharyngotonsillitis (Infections and infestations) | 1/330 | 0/286
Pneumonia (Infections and infestations) | 0/330 | 1/286
Respiratory Syncytial Virus Infection (Infections and infestations) | 0/330 | 1/286
Rhinitis (Infections and infestations) | 7/330 | 7/286
Roseola (Infections and infestations) | 5/330 | 1/286
Sinusitis (Infections and infestations) | 3/330 | 0/286
Skin Infection (Infections and infestations) | 1/330 | 0/286
Tinea Pedis (Infections and infestations) | 0/330 | 1/286
Upper Respiratory Tract Infection (Infections and infestations) | 34/330 | 19/286
Viraemia (Infections and infestations) | 1/330 | 0/286
Viral Infection (Infections and infestations) | 9/330 | 1/286
Viral Pharyngitis (Infections and infestations) | 1/330 | 0/286
Viral Skin Infection (Infections and infestations) | 2/330 | 2/286
Viral upper respiratory tract Infection (Infections and infestations) | 0/330 | 2/286
Arthropod Bite (Injury, poisoning and procedural complications) | 2/330 | 2/286
Arthropod Sting (Injury, poisoning and procedural complications) | 1/330 | 0/286
Contusion (Injury, poisoning and procedural complications) | 1/330 | 0/286
Head Injury (Injury, poisoning and procedural complications) | 1/330 | 0/286
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1/330 | 0/286
Sunburn (Injury, poisoning and procedural complications) | 1/330 | 0/286
Thermal Burn (Injury, poisoning and procedural complications) | 0/330 | 1/286
Anorexia (Metabolism and nutrition disorders) | 2/330 | 1/286
Decreased Appetite (Metabolism and nutrition disorders) | 1/330 | 0/286
Hypervitaminosis A (Metabolism and nutrition disorders) | 1/330 | 0/286
Iron Deficiency (Metabolism and nutrition disorders) | 0/330 | 1/286
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1/330 | 0/286
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1/330 | 0/286
Febrile Convulsion (Nervous system disorders) | 1/330 | 0/286
Headache (Nervous system disorders) | 1/330 | 1/286
Lethargy (Nervous system disorders) | 1/330 | 1/286
Tremor (Nervous system disorders) | 1/330 | 0/286
Crying (Psychiatric disorders) | 1/330 | 0/286
Insomnia (Psychiatric disorders) | 1/330 | 1/286
Restlessness (Psychiatric disorders) | 0/330 | 2/286
Sleep Disorder (Psychiatric disorders) | 0/330 | 1/286
Penile Discharge (Reproductive system and breast disorders) | 0/330 | 1/286
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/330 | 1/286
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1/330 | 2/286
Cough (Respiratory, thoracic and mediastinal disorders) | 15/330 | 9/286
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7/330 | 3/286
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1/330 | 1/286
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1/330 | 0/286
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 3/330 | 2/286
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0/330 | 1/286
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2/330 | 1/286
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 16/330 | 9/286
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2/330 | 1/286
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2/330 | 1/286
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/330 | 1/286
Dermatitis (Skin and subcutaneous tissue disorders) | 1/330 | 0/286
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1/330 | 2/286
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1/330 | 1/286
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1/330 | 0/286
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 26/330 | 9/286
Eczema (Skin and subcutaneous tissue disorders) | 3/330 | 3/286
Erythema (Skin and subcutaneous tissue disorders) | 2/330 | 0/286
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1/330 | 0/286
Rash (Skin and subcutaneous tissue disorders) | 10/330 | 4/286
Rash Macular (Skin and subcutaneous tissue disorders) | 1/330 | 0/286
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1/330 | 0/286
Rash Morbilliform (Skin and subcutaneous tissue disorders) | 8/330 | 1/286
Rash Rubelliform (Skin and subcutaneous tissue disorders) | 1/330 | 0/286
Rash Vesicular (Skin and subcutaneous tissue disorders) | 4/330 | 2/286
Urticaria (Skin and subcutaneous tissue disorders) | 0/330 | 1/286
Bruising, Injection site for VAQTA™ (General disorders) | 6/330 | 7/286
Erythema, Injection site for VAQTA™ (General disorders) | 45/330 | 51/286
Haemorrhage, Injection site for VAQTA™ (General disorders) | 1/330 | 0/286
Nodule, Injection site for VAQTA™ (General disorders) | 1/330 | 0/286
Pain, Injection site for VAQTA™ (General disorders) | 86/330 | 73/286
Rash, Injection site for VAQTA™ (General disorders) | 5/330 | 1/286
Reaction, Injection site for VAQTA™ (General disorders) | 1/330 | 0/286
Swelling, Injection site for VAQTA™ (General disorders) | 32/330 | 38/286
Warmth, Injection site for VAQTA™ (General disorders) | 2/330 | 0/286

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.